CLINICAL TRIAL: NCT02949193
Title: A Phase III Clinical Trial to Investigate the Efficacy and Safety of Evogliptin When Added to Ongoing Metformin Monotherapy in Patients With Type 2 Diabetes
Brief Title: Efficacy and Safety of Evogliptin add-on to Metformin in Patients With type2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA1229_DMC_III
Record Dates: First submitted 2014-02-23; First posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- evogliptin (Experimental): evogliptin 5mg qd add-on to metformin
  Interventions: Drug: evogliptin
- sitagliptin (Active Comparator): sitagliptin 100mg qd add-on to metformin
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: evogliptin — evogliptin 5mg tablet qd + placebo tablet matching to sitagliptin 100mg
  Other Names: Suganon
  Arms: evogliptin
Drug: Sitagliptin — sitagliptin 100 mg tablet qd + placebo tablet matching to evogliptin 5mg
  Other Names: januvia
  Arms: sitagliptin

SUMMARY:
This is a randomized, double-blind, active-controlled, phase III clinical trial to investigate the efficacy and safety of evogliptin when added to ongoing metformin monotherapy in patients with type 2 diabetes who have inadequate glycemic control

DETAILED DESCRIPTION:
1. Evogliptin 5mg Group: Administration with Evogliptin 5mg add-on to metformin for 0-52 weeks.
2. Sitagliptin 100mg Group: Administration with Sitagliptin 100mg add-on to metformin for 0-24 weeks, and with Evogliptin 5mg add-on to metformin for 24-52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with 6.5%≤HbA1c≤11.0% at screening
* Subjects treated with 1,000mg/day or higher dose of metformin for at least 6 weeks prior to screening among people treated with metformin monotherapy for at least 12 weeks before screening
* Subjects with 20kg/m2≤BMI≤40kg/m2 at screening

Exclusion Criteria:

* Subjects with fasting plasma glucose≥270mg/dL at screening
* Patients with type 1 diabetes mellitus, secondary diabetes mellitus or gestational diabetes mellitus
* Subjects with history of myocardial infarction, cerebral infarction within 6 months prior to screening
* Subjects with ALT and AST 2.5 times or higher than upper normal range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2013-05; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
HbA1c | Change from baseline at 24 week
  unit: %

SECONDARY OUTCOMES:
fasting plasma glucose | Change from baseline at 24 week
  unit : mg/dL
HOMA-beta | Change from baseline at 24 week
  unit: %
HbA1c response rate | Change from baseline at 24 weeks
  unit: %

CONTACTS AND LOCATIONS:
Overall Officials: Sung Woo Park, M.D., Ph.D., Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No